CLINICAL TRIAL: NCT02532231
Title: PD-1 Inhibition With Nivolumab for the Treatment of Patients With Acute Myeloid Leukemia in Remission at High Risk for Relapse
Brief Title: Nivolumab in AML in Remission at High Risk for Relapse
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-0213; NCI-2015-01522 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2015-0213 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2015-08-21; First posted 2015-08-25 (Estimated); Results first posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Acute Myeloid Leukemia Arising From Previous Myelodysplastic Syndrome; Adult Acute Myeloid Leukemia in Remission; Blasts Under 10 Percent of Bone Marrow Nucleated Cells; Therapy-Related Myeloid Neoplasm
MeSH Terms: interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (nivolumab) (Experimental): Patients receive nivolumab IV over 1 hour on days 1 and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. After cycle 6, patients may receive nivolumab on day 1 only. After cycle 12, patients may receive nivolumab on day 1 of every 3 cycles. Patients experiencing disease progression may go back to receiving treatment on days 1 and 15 of each cycle.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Nivolumab

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo

SUMMARY:
This phase II trial studies how well nivolumab works in treating patients with acute myeloid leukemia that has decreased or disappeared but may still be in the body (remission), and is at high risk for returning (relapse). Immunotherapy with monoclonal antibodies, such as nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the anti-leukemic effects of nivolumab in patients with acute myeloid leukemia (AML) who have achieved a 1st complete remission (CR) after induction chemotherapy and consolidation chemotherapy and have high risk for relapse, or have achieved a 2nd CR.

SECONDARY OBJECTIVES:

I. To evaluate the immunologic responses to nivolumab among patients with AML in CR status post standard chemotherapy.

II. To determine whether response to nivolumab correlates with immunologic responses.

III. To evaluate assessment of minimal residual disease (MRD) by flow cytometry as a predictor of response to immune therapy in treatment of AML and changes during the course of therapy with nivolumab.

IV. To evaluate time to relapse and overall survival. V. To evaluate the toxicity profile of nivolumab among patients with AML in CR.

OUTLINE:

Patients receive nivolumab intravenously (IV) over 1 hour on days 1 and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. After cycle 6, patients may receive nivolumab on day 1 only. After cycle 12, patients may receive nivolumab on day 1 of every 3 cycles. Patients experiencing disease progression may go back to receiving treatment on days 1 and 15 of each cycle.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients with AML in remission (defined as CR, CR with incomplete platelet recovery -CRp-, CR with incomplete hematologic recovery -CRi-, or partial remission defined as a bone marrow with < 10% blasts after therapy with or without hematologic recovery)
* High risk for relapse defined as: 1st CR with high risk features for relapse (including history of prior malignancy treated with chemotherapy or radiotherapy, or history of myelodysplastic syndrome, myeloproliferative disorder, chronic myelomonocytic leukemia, myelodysplastic syndrome [MDS]/myeloproliferative neoplasm [MPN] or other hematologic malignancy thought to have evolved to AML [i.e., secondary AML, (sAML)]; high risk cytogenetics at diagnosis; fms-related tyrosine kinase 3 [FLT3] mutated at diagnosis; or presence or minimal residual disease assessed by polymerase chain reaction [PCR], cytogenetics, and/or flow cytometry at time of enrollment) 2nd CR regardless of disease characteristics at the time of diagnosis
* Have received induction chemotherapy and at least one cycle of consolidation chemotherapy; patients should have achieved a CR within 12 months of enrollment onto protocol
* No further chemotherapy or stem cell transplant (SCT) planned at the time of enrollment
* Creatinine =< 1.5 x upper limit of normal (ULN)
* Serum bilirubin =< 1.5 x ULN
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x ULN
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Females of childbearing potential must have a negative serum or urine beta human chorionic gonadotropin (b-hCG) pregnancy test result within 24 hours prior to the first dose of treatment and must agree to use an effective contraception method during the study and for 23 weeks after the last dose of the study drug; females of non-childbearing potential are those who are postmenopausal greater than 1 year or who have had a bilateral tubal ligation or hysterectomy
* Males who have partners of childbearing potential must agree to use an effective contraceptive method during the study and for 31 weeks following the last dose of study drug
* Patients or their legally authorized representative must provide written informed consent

Exclusion Criteria:

* History of another primary invasive malignancy that has not been definitively treated or in remission for at least 2 years; patients with non-melanoma skin cancers or with carcinomas in situ are eligible regardless of the time from diagnosis (including concomitant diagnoses)
* Any major surgery, radiotherapy, chemotherapy, biologic therapy, immunotherapy, experimental therapy within 2 weeks prior to the first dose of the study drugs
* Patients with any other known concurrent severe and/or uncontrolled medical condition (e.g. uncontrolled diabetes; cardiovascular disease including congestive heart failure New York Heart Association [NYHA] class III or IV, myocardial infarction within 6 months, and poorly controlled hypertension; chronic renal failure; or active uncontrolled infection) which, in the opinion of the investigator could compromise participation in the study
* Patients unwilling or unable to comply with the protocol
* Patients who are on steroids (> 10 mg/day or equivalent) or immune suppression medications
* Patients with autoimmune diseases (e.g., rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, autoimmune vasculitis [e.g., Wegener's granulomatosis])
* Patients with a history of inflammatory bowel disease such as Crohn's disease and ulcerative colitis
* Patients known to be positive for hepatitis B surface antigen expression or with active hepatitis C infection (positive by polymerase chain reaction or on antiviral therapy for hepatitis C within the last 6 months), or with known human immunodeficiency virus (HIV) infection
* Current therapy with other systemic anti-neoplastic or anti-neoplastic investigational agents
* Females who are pregnant or lactating
* Patients with history of previous immunomodulatory therapy (not including lenalidomide or thalidomide)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-10-19 (Actual); Primary Completion 2023-08-08 (Actual); Study Completion 2023-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tapan M Kadia, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Shallis RM, Podoltsev NA. Maintenance therapy for acute myeloid leukemia: sustaining the pursuit for sustained remission. Curr Opin Hematol. 2021 Mar 1;28(2):110-121. doi: 10.1097/MOH.0000000000000637. PMID 33394722
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Nivolumab)
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Nivolumab)
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 3
Age, Continuous [Median (Full Range); unit: years] | 56 [31 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 10
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Recurrence-free Survival Rate
Description: Time from date of treatment start until the date of first objective documentation of disease-relapse.
Time Frame: Up to 7 years 9 months
Measure: Median (Full Range); unit: Months
Arm/Group | Treatment (Nivolumab)
Number analyzed (Participants) | 15
Months | 8.5 [1 to 47]

2. Secondary Outcome: Number of Participants With Immunologic Responses to Nivolumab Among Patients With Acute Myeloid Leukemia (AML) in Complete Remission (CR) Status Post Standard Chemotherapy
Description: Participants with Immunologic responses to nivolumab among patients with acute myeloid leukemia (AML) in complete remission (CR) status post standard chemotherapy. CR is Neutrophil count >/= 1.0 x 10^9/L, with a platelet count of >/+ x 10 ^ 9/L
Time Frame: Every 2 cycles (+/-1 cycle) for the first 6 cycles, then every 3 months while on study, then as clinically indicated till relapse; up to 7 years, 9 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Nivolumab)
Number analyzed (Participants) | 15
Participants | 6

3. Secondary Outcome: Number of Participants Who Changed From MRD Postive to MRD Negative During Therapy With Nibolumab
Description: Assessed by flow cytometry as a predictor of response to immune therapy in treatment of AML. The number of participants who were MRD Positive at the start of therapy with nivolumab and changed to MRD Negative during treatment.
Time Frame: as for outcome 2
Population: There were 6 participants who were MRD negative and 9 who were MRD positive at the beginning of therapy with nivolumab. Therefor the number of participants analyzed for this outcome were 9 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Nivolumab)
Number analyzed (Participants) | 9
Participants | 2

4. Secondary Outcome: Time to Relapse
Description: Time from date of treatment start until the date of first objective documentation of disease-relapse.
Time Frame: Up to 7 years 9 months
Measure: Median (Full Range); unit: Months
Arm/Group | Treatment (Nivolumab)
Number analyzed (Participants) | 9
Months | 2 [1 to 9]

5. Secondary Outcome: Overall Survival
Description: Time from date of treatment start until date of death due to any cause or last Follow-up.
Time Frame: Up to 7 years 9 months
Measure: Median (Full Range); unit: Months
Arm/Group | Treatment (Nivolumab)
Number analyzed (Participants) | 15
Months | NA [2 to 47] — At the time of study termination the median overall survival was not reached.

ADVERSE EVENTS:
Time Frame: Up to 7 years 9 months
Arm/Group | Treatment (Nivolumab)
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 6/15
Other Adverse Events (participants affected / at risk) | 8/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Nivolumab) (N=15)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Acute Coronary Syndrome (Cardiac disorders) | 1 (1)
Back Pain (General disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 2 (2)
Fracture (Injury, poisoning and procedural complications) | 1 (2)
Hypotension (Vascular disorders) | 1 (2)
Infection (Infections and infestations) | 1 (1)
Lung Infection (Infections and infestations) | 3 (5)
Nausea (Gastrointestinal disorders) | 1 (1)
Otitis Externa (Ear and labyrinth disorders) | 1 (1)
Papulopustular Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (2)
Upper Respiratory Infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Nivolumab) (N=15)
Skin Lesions-Itchy (Skin and subcutaneous tissue disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Thyroid function, low (hypothyroidism) (Endocrine disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
AST, SGOT (serum glutamic oxaloacetic transaminase) (Investigations) | 1 (1)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1 (1)
Pain--Select (General disorders) | 2 (3)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1 (1)
Distension/bloating, abdominal (Gastrointestinal disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Febrile neutropenia (Infections and infestations) | 1 (1)
Mucositis/stomatitis (clinical exam) (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-09): https://cdn.clinicaltrials.gov/large-docs/31/NCT02532231/Prot_SAP_000.pdf